CLINICAL TRIAL: NCT06525701
Title: Surgeon Core-strengthening Program as a Modifier for Exertion Associated With Vaginal Surgery: the SCORE Randomized Controlled Trial
Brief Title: Surgeon Core-strengthening Program as a Modifier for Exertion Associated With Vaginal Surgery
Acronym: SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Marian G. Acevedo Alvarez, PI, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 218292
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Injury
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The intervention group will complete a core workout lasting 20 minutes twice a week for 4 weeks
Who Masked: Investigator
Masking Description: The control group will not have an exercise regimen. The PI will be blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants randomized to the exercise group will be asked to perform the SCORE workout two times each week for 4 weeks prior to their urogynecology rotation and for 4 weeks during the rotation.
  Interventions: Other: Execise Group; Other: Control Group
- Control Group (Active Comparator): No additional exercises or tasks are requested of control participants. Control group participants will perform or not perform exercise as they otherwise would outside of the study
  Interventions: Other: Execise Group; Other: Control Group

INTERVENTIONS:
Other: Execise Group — SCORE workout: eight exercises done sequentially: bicycles, balancing dog, windshield wipers, three-point plank, kayaker, super push-ups, bridge, and side plank. These workouts are modified from the core regimen recommended by Steve House and Scott Johnston in their book Training for the New Alpinism: A Manual for the Climber as Athlete (House 2014). Each exercise is done until fatigue: when the individual is no longer able to complete the exercise with good form. The participant then rests for approximately thirty to sixty seconds before beginning the next exercise. Passive stretching can be performed during the rest periods. The workout is complete at twenty minutes. Those individuals who complete all eight exercises in less than twenty minutes begin again with the first exercise (bicycles) and continue until reaching twenty minutes. The workout is thus adaptive-seamlessly increasing in repetitions as an individual's strength and endurance increase.
Other: Control Group — No additional exercises or tasks are requested of control participants. Control group participants will perform or not perform exercise as they otherwise would outside of the study.

SUMMARY:
Work-related musculoskeletal pain and injury is a growing concern in surgery. Vaginal surgery has unique ergonomic risks, but no studies have addressed the potential for an exercise regimen to reduce physical strain by vaginal surgeons

DETAILED DESCRIPTION:
Surgical ergonomics is a burgeoning field, spurred by the recognition of the high prevalence of work-related musculoskeletal pain and injury in practicing surgeons including obstetrician/gynecologists. Surgery is often a demanding physical task, and the muscles and joints that are stressed vary by the surgical approach. Vaginal surgery has unique ergonomic challenges, particularly for assistants who may need to laterally bend their torsos to visualize the surgical field while still holding retractors. This is often a compromising physical position for the back, the shoulders, and sometimes the neck which increases the risk of acute or chronic musculoskeletal injury. The risk of injury can be thought of as a discrepancy between the demands of the task and the individual's physical capabilities. Surgeons' injury risk may be decreased if their physical capabilities can be improved through exercise. Most existing publications on surgical ergonomics have focused on raising awareness and on environmental changes such as optimizing surgeon posture during the case or introducing micro-breaks and stretching. Few publications have assessed a structured exercise program with the goal of decreasing surgeon pain or fatigue during and after surgery. To our knowledge, no studies have addressed this in vaginal surgery.

ELIGIBILITY:
Inclusion Criteria:

Participant: ob/gyn resident or urology resident or urogyn fellow or urogyn attending Case: vaginal prolapse surgery >2 hours in length

Exclusion Criteria:

Participant:

1. Actively in physical therapy
2. Joint surgery or joint injury within last 12 weeks
3. Pregnant
4. Less than 6 weeks postpartum

Case:

1. Vaginal surgery <2 hours in length
2. Non-prolapse vaginal surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The effect of a core-strengthening program on surgeons' physical exertion during and after vaginal prolapse surgery using the Borg rating of perceived exertion (Borg CR10). To determine the effect of a core-strengthening program on surgeon | 8-12 weeks
  The effect of a core-strengthening program on surgeons' physical exertion during and after vaginal prolapse surgery as measured by the Borg Category Ratio (CR-10). The Borg Category Ratio scale is a self-reported tool that describes level of exertion and ranges from 0-10 where larger numbers represent greater exertion.

SECONDARY OUTCOMES:
To describe the baseline core strength in a population of vaginal surgeons using the validated Core Score | 8-12 weeks
  • Core Score: The Core Score ranges from 0-12 where higher scores indicate better performance on core-related exercises.
To describe the execise habits and activity level in a populationa of vaginal surgeons using activity tracker data and the International Physical Activity Questionnaire. | 8-12 weeks
  • International Physical Activity Questionnaire-Short Form (IPAQ-SF): Participant responses on time spent walking, doing moderate exercise, and doing vigorous exercise are first compared to a rubric for the categorical score. The categorical score ranges 1-3 where 1 is "inactive" and 3 is "health-enhancing physical activity". Participant responses are also used to calculate the weekly metabolic equivalent (MET) minutes where a higher number indicates more time spent being physically active.
To measure the effect of a core-strengthening program on surgeons' pain during and after vaginal prolapse surgery using the PROMIS Pain Intensity-Short Form (PI-SF) and body diagrams. | 8-12 weeks
  • PROMIS Pain Intensity-Short Form (PI-SF): The raw score ranges from 3-15 where higher scores indicate more pain. Raw scores are converted to t-scores where a t-score of 50 represents the average in the United States population.
To measure objective and subjective change in core strength after completion of the core-strengthening program using the Core Score and Patient Global Impression of Improvement (PGI-I). | 8-12 weeks
  • Patient Global Impression of Improvement (PGI-I): Lower Patient Global Impression of Improvement scores indicate more improvement. PGI-I ranges from 1 ("very much better") to 7 ("very much worse").

CONTACTS AND LOCATIONS:
Overall Officials: Marian Acevedo-Alvarez, MD, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giagio S, Volpe G, Pillastrini P, Gasparre G, Frizziero A, Squizzato F. A Preventive Program for Work-related Musculoskeletal Disorders Among Surgeons: Outcomes of a Randomized Controlled Clinical Trial. Ann Surg. 2019 Dec;270(6):969-975. doi: 10.1097/SLA.0000000000003199. PMID 30672801
- [Background] Allespach H, Sussman M, Bolanos J, Atri E, Schulman CI. Practice Longer and Stronger: Maximizing the Physical Well-Being of Surgical Residents with Targeted Ergonomics Training. J Surg Educ. 2020 Sep-Oct;77(5):1024-1027. doi: 10.1016/j.jsurg.2020.04.001. Epub 2020 Aug 4. PMID 32763097
- [Background] Al Reshidi FS. Level of Physical Activity of Physicians Among Residency Training Program At Prince Sultan Military Medical City, Riyadh, KSA 2014. Int J Health Sci (Qassim). 2016 Jan;10(1):39-47. doi: 10.12816/0031215. PMID 27004056
- [Background] Bertolaccini L, Viti A, Terzi A. Ergon-trial: ergonomic evaluation of single-port access versus three-port access video-assisted thoracic surgery. Surg Endosc. 2015 Oct;29(10):2934-40. doi: 10.1007/s00464-014-4024-6. Epub 2014 Dec 17. PMID 25515979
- [Background] Cruz-Montecinos C, Bustamante A, Candia-Gonzalez M, Gonzalez-Bravo C, Gallardo-Molina P, Andersen LL, Calatayud J. Perceived physical exertion is a good indicator of neuromuscular fatigue for the core muscles. J Electromyogr Kinesiol. 2019 Dec;49:102360. doi: 10.1016/j.jelekin.2019.102360. Epub 2019 Sep 28. PMID 31580987
- [Background] Choi SH, Kuchta K, Rojas A, Mehdi SA, Ramirez Barriga M, Hays S, Talamonti MS, Hogg ME. Residents perform better technically, have less stress and workload, and prefer robotic to laparoscopic technique during inanimate simulation. Surg Endosc. 2023 Sep;37(9):7230-7237. doi: 10.1007/s00464-023-10216-5. Epub 2023 Jul 3. PMID 37395804
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Dairywala MI, Gupta S, Salna M, Nguyen TC. Surgeon Strength: Ergonomics and Strength Training in Cardiothoracic Surgery. Semin Thorac Cardiovasc Surg. 2022 Winter;34(4):1220-1229. doi: 10.1053/j.semtcvs.2021.09.015. Epub 2021 Sep 29. PMID 34597795
- [Background] Friedrich J, Brakke R, Akuthota V, Sullivan W. Reliability and Practicality of the Core Score: Four Dynamic Core Stability Tests Performed in a Physician Office Setting. Clin J Sport Med. 2017 Jul;27(4):409-414. doi: 10.1097/JSM.0000000000000366. PMID 28653966
- [Background] Henriksen A, Haugen Mikalsen M, Woldaregay AZ, Muzny M, Hartvigsen G, Hopstock LA, Grimsgaard S. Using Fitness Trackers and Smartwatches to Measure Physical Activity in Research: Analysis of Consumer Wrist-Worn Wearables. J Med Internet Res. 2018 Mar 22;20(3):e110. doi: 10.2196/jmir.9157. PMID 29567635
- [Background] Jo D, Bilodeau M. Rating of perceived exertion (RPE) in studies of fatigue-induced postural control alterations in healthy adults: Scoping review of quantitative evidence. Gait Posture. 2021 Oct;90:167-178. doi: 10.1016/j.gaitpost.2021.08.015. Epub 2021 Aug 25. PMID 34492503
- [Background] Keohane DM, McGillivary NA, Daly B. Physical activity levels and perceived barriers to exercise participation in Irish General Practitioners and General Practice trainees. Ir Med J. 2018 Feb 9;111(2):690. PMID 29952439
- [Background] Kopkash K, Novak K, Murphy R, Deliere A, Kuchta K, Rabbitt S, Pesce C, Winchester D, Yao K. Improving the Breast Surgeon's Ergonomic Workload for Nipple-Sparing Mastectomies Using Exercise and Operating Room Positioning Protocol. Ann Surg Oncol. 2021 Oct;28(10):5698-5706. doi: 10.1245/s10434-021-10447-7. Epub 2021 Jul 27. PMID 34318384
- [Background] Kromberg LS, Kildebro NV, Mortensen LQ, Amirian I, Rosenberg J. Microbreaks in Laparoscopic Appendectomy have No Effect on Surgeons' Performance and Well-being. J Surg Res. 2020 Jul;251:1-5. doi: 10.1016/j.jss.2020.01.007. Epub 2020 Feb 21. PMID 32092608
- [Background] Lentz TA, Rhon DI, George SZ. Predicting Opioid Use, Increased Health Care Utilization and High Costs for Musculoskeletal Pain: What Factors Mediate Pain Intensity and Disability? J Pain. 2020 Jan-Feb;21(1-2):135-145. doi: 10.1016/j.jpain.2019.06.004. Epub 2019 Jun 13. PMID 31201989
- [Background] Meltzer AJ, Hallbeck MS, Morrow MM, Lowndes BR, Davila VJ, Stone WM, Money SR. Measuring Ergonomic Risk in Operating Surgeons by Using Wearable Technology. JAMA Surg. 2020 May 1;155(5):444-446. doi: 10.1001/jamasurg.2019.6384. PMID 32159745
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Parry DA, Oeppen RS, Amin MSA, Brennan PA. Could exercise improve mental health and cognitive skills for surgeons and other healthcare professionals? Br J Oral Maxillofac Surg. 2018 Jun;56(5):367-370. doi: 10.1016/j.bjoms.2018.03.005. Epub 2018 Apr 9. PMID 29650472
- [Background] Rodrigues H, Cobucci R, Oliveira A, Cabral JV, Medeiros L, Gurgel K, Souza T, Goncalves AK. Burnout syndrome among medical residents: A systematic review and meta-analysis. PLoS One. 2018 Nov 12;13(11):e0206840. doi: 10.1371/journal.pone.0206840. eCollection 2018. PMID 30418984
- [Background] Selvaraj CS, Abdullah N. Physically active primary care doctors are more likely to offer exercise counselling to patients with cardiovascular diseases: a cross-sectional study. BMC Prim Care. 2022 Mar 29;23(1):59. doi: 10.1186/s12875-022-01657-3. PMID 35350999
- [Background] Stone AA, Broderick JE, Junghaenel DU, Schneider S, Schwartz JE. PROMIS fatigue, pain intensity, pain interference, pain behavior, physical function, depression, anxiety, and anger scales demonstrate ecological validity. J Clin Epidemiol. 2016 Jun;74:194-206. doi: 10.1016/j.jclinepi.2015.08.029. Epub 2015 Nov 25. PMID 26628334
- [Background] Suija K, Pechter U, Maaroos J, Kalda R, Ratsep A, Oona M, Maaroos HI. Physical activity of Estonian family doctors and their counselling for a healthy lifestyle: a cross-sectional study. BMC Fam Pract. 2010 Jun 18;11:48. doi: 10.1186/1471-2296-11-48. PMID 20565892
- [Background] Whittaker RL, Sonne MW, Potvin JR. Ratings of perceived fatigue predict fatigue induced declines in muscle strength during tasks with different distributions of effort and recovery. J Electromyogr Kinesiol. 2019 Aug;47:88-95. doi: 10.1016/j.jelekin.2019.05.012. Epub 2019 May 18. PMID 31136944
- [Background] Winters JN, Sommer NZ, Romanelli MR, Marschik C, Hulcher L, Cutler BJ. Stretching and Strength Training to Improve Postural Ergonomics and Endurance in the Operating Room. Plast Reconstr Surg Glob Open. 2020 May 13;8(5):e2810. doi: 10.1097/GOX.0000000000002810. eCollection 2020 May. PMID 33133890
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Yurteri-Kaplan LA, Park AJ. Surgical Ergonomics and Preventing Work-Related Musculoskeletal Disorders. Obstet Gynecol. 2023 Mar 1;141(3):455-462. doi: 10.1097/AOG.0000000000005079. Epub 2023 Feb 2. No abstract available. PMID 36735407